CLINICAL TRIAL: NCT02606643
Title: Balloon Catheter for Cervical Ripening With or Without Traction: A Randomized Controlled Trial
Brief Title: Balloon Catheter for Cervical Ripening
Acronym: 25148
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: StLouisU
Record Dates: First submitted 2015-08-24; First posted 2015-11-17 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-02

CONDITIONS: Cervical Dilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Catheter to slight traction (Active Comparator): For the "Tension" arm (research related), slight tension will be placed on the catheter, which will then be taped to the patient's inner thigh. The tension will be assessed and retaped as needed every 30 minutes by the research and/or the nursing staff.
  Only slight tension will be applied to those catheters assign to the tension group. The catheter will be taped to the inner thigh so there is no "sag" in the catheter from the urethra to the tape. There is no method or device to "measure" the tension placed on these catheters, if the patient moves her leg it can lessen or increase the tension, these are known factors.
  Interventions: Procedure: Slight traction
- Group 2 Catheter to no traction (Active Comparator): Foley catheter to no traction placed as SOC "No traction" applied
  Interventions: Procedure: Foley Catheter to no traction

INTERVENTIONS:
Procedure: Slight traction — Slight traction will be applied to the balloon catheter
  Arms: Group 1 Catheter to slight traction
Procedure: Foley Catheter to no traction — Foley Catheter to no traction
  Arms: Group 2 Catheter to no traction

SUMMARY:
Once admitted, women who will have a transcervical balloon catheter inserted for induction will be approached for participation in this study. If they agree to be take part in this study (tape or no tape) they will be randomized into the study. After the balloon catheter is inserted, the balloon will then be filled with approximately 50-60 mL of normal saline, this is normal procedure.

Study related: If randomized to "No Taping" the foley will be positioned comfortable and not placed to tension. For the "Tension" arm, tension will be placed on the balloon catheter, which will then be taped to the patient's inner thigh. The tension will be assessed and retaped as needed approximately every 30 minutes by the research and/or the nursing staff.

DETAILED DESCRIPTION:
Once admitted, women who are schedule for induction and who's physician has order a balloon catheter, they will have a transcervical balloon catheter inserted-this is normal care. Patients will be placed in the dorsal lithotomy position in the delivery bed. The cervix will be examined digitally (this is the standard of care). The balloon catheter will be inserted by feel and passed through the cervix until the balloon is above the internal os. The balloon will then filled with approximately 50-60 mL of normal saline. This procedure is standard of care.

Randomization: 63 cards will be prepared to read "tape for tension" and 63 will be prepared to read "No tape/No Tension". These cards will be sealed in opaque envelopes and kept in the PI's office. After consent is obtained the PI will be notified and a sealed envelope will be opened and the patient and staff will be notified.

If randomized to "No tension" the catheter will be positioned comfortable and not placed to tension (this is currently the standard at SSM - Saint Mary's Hospital ).

For the "Tension" arm (research related), slight tension will be placed on the catheter, which will then be taped to the patient's inner thigh. The tension will be assessed and retaped as needed every 30 minutes by the research and/or the nursing staff.

Only slight tension will be applied to those catheters assign to the tension group. The catheter will be taped to the inner thigh so there is no "sag" in the catheter from the urethra to the tape. There is no method or device to "measure" the tension placed on these catheters, if the patient moves her leg it can lessen or increase the tension, these are known factors.

As part of the induction process, patients will be started on an infusion of oxytocin, this is the practice at SSMHC, unless there is a reason not to use oxytocin such as nonreassuring fetal heart tracing. In this situation it is the physician's choice of what to use for induction. Oxytocin is initiated at 2 milliunits/minute and increased 1-2 milliunits/minute approximately every 20 minutes to a maximum of 6 milliunits/minute while the Foley is in place.

After expulsion of the balloon, the resident or attending physician will performed a cervical examination to document the time and the cervical examination, and the oxytocin will be titrated to achieve acceptable contraction rates without tachysystole -this is standard care.

The patient's labor and delivery will be managed according to routine obstetric and institutional protocols. All patients will have continuous fetal heart rate and uterine activity monitoring.

Chart review will be performed on both the maternal and infant medical record from admission to discharge.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestation
* Bishop score less than or equal to 6
* cephalic presentation

Exclusion Criteria:

* prostaglandins given this admission
* any medical conditions precluding vaginal delivery
* significant cervical or intrauterine infection
* significant vaginal bleeding
* intrauterine fetal demise
* low lying placenta
* prior cervical surgery
* latex allergy

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Fruhman, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Catheter to Slight Traction: 68 patients were analyzed in the tension group
- Group 2 Catheter to no Traction: 76 patients were analyzed in the no tension group
Period: Overall Study
Arm/Group | Group 1 Catheter to Slight Traction | Group 2 Catheter to no Traction
Started | 68 | 76
Completed | 67 | 73
Not Completed | 1 | 3
Not completed — did not meet inclusion criteria | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Catheter to Slight Traction: Once the decision was made to use a transcervical catheter and the patient was not in labor, the patient was approached. After informed consent was obtained from each participant, an 18 French 30 cc Foley bulb was placed digitally by the housestaff, with or without a stylette. The balloon was filled with 50 cc of saline as this is the standard at our institution. Patients randomized to tension had their catheter taped with applied tension to the inner thigh. Tension was replaced approximately every 30 minutes as needed. If the catheter was not expelled after12 hours, the balloon was deflated and the catheter was removed.
- Group 2 Catheter to no Traction: Once the decision was made to use a transcervical catheter and the patient was not in labor, the patient was approached. After informed consent was obtained from each participant, an 18 French 30 cc Foley bulb was placed digitally by the housestaff, with or without a stylette. The balloon was filled with 50 cc of saline as this is the standard at our institution. Patients randomized to no tension did not have any tension applied to their catheter. After randomization clinicians were not blinded to the allocated group. If the catheter was not expelled after12 hours, the balloon was deflated and the catheter was removed.
- Total: Total of all reporting groups
Arm/Group | Group 1 Catheter to Slight Traction | Group 2 Catheter to no Traction | Total
Number analyzed (Participants) | 68 | 76 | 144
Age, Continuous [Mean (Full Range); unit: years] | 26 [23 to 30] | 26 [22 to 30] | 026 [22 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 76 | 144
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — 11 participants failed screening and were not included in analysis
  participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 41 | 53 | 94
    White | 20 | 17 | 37
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 68 | 76 | 144
Gestational age at enrollment (wk [Mean (Full Range); unit: weeks] | 39.1 [37.6 to 40.4] | 39.0 [37.6 to 40.1] | 39.05 [37.6 to 40.1]
Body mass index at admission [Mean (Full Range); unit: kg/m2] — Body mass index at admission (kg/m^2)
  kg/m2 | 33.1 [28.9 to 41.6] | 37.0 [29.0 to 42.2] | 35.05 [28.9 to 42.2]
Bishop score at time of transcervical [Mean (Full Range); unit: units on a scale] — A women with a low score of 1 would not expected go into labor for about 3 weeks. A woman with a higher score score of 10 could be expected to go into labor within a few days.
  units on a scale | 4 [3 to 5] | 3.5 [3 to 5] | 3.75 [3 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Duration
Description: Hours of labor
Time Frame: hours to delivery 0-26
Population: an alpha level of .05, and a level of power of 80%. These parameters required a sample size of 63 patients per group
Measure: Mean (Full Range); unit: hours
Groups:
- Group 1 Slight Tension: Patients randomized to tension had their catheter taped with applied tension to the inner thigh. Tension was replaced approximately every 30 minutes as needed.
- Group 2 no Tension: Patients randomized to no tension did not have any tension applied to their catheter.
Arm/Group | Group 1 Slight Tension | Group 2 no Tension
Number analyzed (Participants) | 67 | 73
hours | 16.2 [12.6 to 23.5] | 16.9 [12.4 to 25.6]
Statistical Analysis 1: Comparison: Group 1 Slight Tension vs Group 2 no Tension; an alpha level of .05, and a level of power of 80%. These parameters required a sample size of 63 patients per group; Test type: Superiority or Other; p = 0.814, Chi-squared

2. Secondary Outcome: Deliveries Via Cesarean Delivery
Description: What number of deliveries in the tension and no tension groups were via Cesarean delivery
Time Frame: intraoperative
Measure: Number; unit: participants
Groups:
- Group 1 Slight Tension; Group 2 no Tension: Number of Cesarean deliveries in the no tension group
Arm/Group | Group 1 Slight Tension | Group 2 no Tension
Number analyzed (Participants) | 67 | 73
participants | 17 | 27

3. Secondary Outcome: Vaginal Delivery Within 24 Hours
Description: vaginal delivery within 24 hours-not all deliveries were within 24hours
Time Frame: 24 hours
Population: Twenty four hour Vaginal delivery between groups
Measure: Number; unit: participants
Groups:
- Delivery Within 24 Hours; Group 2 no Tension: The primary and secondary outcome data were not normally distributed. Therefore, medians and interquartile ranges are reported and compared. Means and standard deviations for the primary outcome were included in order to facilitate comparisons to other published research.
Arm/Group | Delivery Within 24 Hours | Group 2 no Tension
Number analyzed (Participants) | 52 | 52
participants | 41 | 37

ADVERSE EVENTS:
Time Frame: 6 months post delivery
Groups:
- Group 1: Slight Tension
- Group 2: no Tension
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/73
Other Adverse Events (participants affected / at risk) | 0/67 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No